CLINICAL TRIAL: NCT06702995
Title: A Phase Ib/II Study of XNW5004 Tablet in Combination With Enzalutamide in Subjects With Metastatic Castration-resistant Prostate Cancer (mCRPC) Who Failed Prior Novel Hormone Therapy
Brief Title: Study of XNW5004 Tablet in Combination With Enzalutamide in Subjects With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XNW5004-Ib/II-01
Record Dates: First submitted 2024-11-11; First posted 2024-11-25 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer; mCRPC (Metastatic Castration-resistant Prostate Cancer)
Keywords: XNW5004; Enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase Ib (Experimental): Participants with mCRPC will receive XNW5004 at escalating dose levels in combination with enzalutamide.
  Interventions: Drug: XNW5004; Drug: enzalutamide
- Phase IIa (Experimental): Participants with mCRPC will receive XNW5004 in combination with enzalutamide.
  Interventions: Drug: XNW5004; Drug: enzalutamide
- Phase IIb (Experimental): Participants with mCRPC will receive XNW5004 in combination with enzalutamide or enzalutamide alone
  Interventions: Drug: XNW5004; Drug: enzalutamide

INTERVENTIONS:
Drug: XNW5004 — Oral continuous
  Other Names: EZH2i
Drug: enzalutamide — enzalutamide 160 mg (four 40 mg capsules) orally once daily
  Other Names: Xtandi

SUMMARY:
In this phase Ib/II study, participants with metastatic castration-resistant prostate cancer (mCRPC) who failed prior novel hormone therapy will be treated with XNW5004 in combination with enzalutamide.

DETAILED DESCRIPTION:
This is a multicenter, phase Ib/II clinical trial, divided into three parts:

The part1 is the dose escalation study of XNW5004 combined with Enzalutamide (Dose escalation in phase Ib) .

The part2 is the dose expansion study of XNW5004 combined with Enzalutamide (Dose expansion in phase IIa).

The phase Ib and IIa will evaluate the safety, tolerability and preliminary anti-tumor activity of XNW5004 in combination with enzalutamide to determine the recommended phase II dose (RP2D).

The part3 is an open label, randomized phase 2 study (Phase IIb). The patients with mCRPC will be enrolled to assess the efficacy of XNW5004 at the RP2D in combination with Enzalutamide in comparison with Enzalutamide alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign an approved informed consent form (ICF).
* Age at the time of consent ≥ 18 years;
* Life expectancy of ≥ 3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
* Prostate adenocarcinoma confirmed by histological or cytological examination, except neuroendocrine carcinoma or small cell carcinoma;
* Metastatic prostate cancer disease, documented by CT/MRI imaging/bone scan ;
* Ongoing luteinizing hormone-releasing hormone agonist (LHRHa) or antagonist therapy (medical castration) or prior bilateral orchiectomy (surgical castration); subjects who have not undergone bilateral orchiectomy must be scheduled for Maintain effective LHRHa therapy throughout the study period;
* Testosterone at castration level (≤50ng/dL or 1.7nmol/L) at screening;
* Progressive disease in the setting of medical or surgical castration for study entry, the subject has 1 or more of the following 3 items: (1) PSA progression, defined as PSA > 1ng/ml and at least 2 episodes of PSA level elevation ≥ 1 week apart; (2) disease progression as defined by RECIST 1.1; (3) bone disease progression as defined by PCWG3 criteria, i.e., ≥ more than 2 new lesions found on bone scan;
* Previous anti-tumor therapy meet the following conditions： Ib and IIb: Failure of previous abiraterone acetate therapy (refers to disease progression during abiraterone acetate treatment; disease progression is defined as the same as in Article 9 of the enrollment criteria), and no next generation androgen receptor inhibitors (enzalutamide or apalutamide, etc.) have been used; IIb: Failure of previous only one approved novel hormone therapy, such as abiraterone acetate, apalutamide, darolutamide and rezvilutamide, etc., except enzalutamide；
* Adequate hematologic and non-hematologic function during the screening.
* Must agree to take adequate contraceptive measures from the beginning of the study to at least 3 months after the last dose of the test drug, and prohibit sperm donation;
* Ability to comply with all procedures of the clinical trial protocol.

Exclusion Criteria:

* Previous anti-tumor therapy meet the following conditions： Ib and IIb: previously received any next generation androgen receptor antagonists (such as enzalutamide, apalutamide, proxalutamide and rezvilutamide, etc.) ； IIa: previously received with enzalutamide or more than 1 novel hormone therapy;
* Prior chemotherapy for castration resistant disease (including but not limited to ADCs);
* Prior exposure to EZH2 inhibitor(s) (including but not limited to tazemetostat and EZH1/2 inhibitors);
* Subjects who received anti-tumor therapies including chemotherapy, immunotherapy, radical radiotherapy, major surgery, targeting therapy and other anti-tumor therapies within 4 weeks or 5 half-lives of the drug (whichever is shorter) before the first dose; or received palliative radiotherapy within 2 weeks before the first dose;
* Plan to receive any other anti-tumor therapy during this trial;
* Subjects who participated in any other clinical trial of anti-tumor therapy within 28 days before the first dosing, and the last dose of other anti-tumor trial drug is within 28 days prior to the first administration of study drug in this trial;
* Central nervous system metastasis or disease;
* Severe bone injury caused by tumor bone metastasis judged by the investigator, including severe bone pain with poor control, pathological fractures of important sites and spinal cord compression that occurred in the past 6 months or are expected to occur in the near future, etc.;
* Subjects who have a history of other malignancies within 3 years prior to enrollment and do not meet the criteria for clinical cure. This exclusion criterion does not apply to skin basal cell carcinoma or squamous cell carcinoma with local treatment methods available and has been cured, superficial bladder cancer, intraductal breast carcinoma in situ, and papillary thyroid carcinoma;
* Subjects who experienced stroke or other serious cerebrovascular diseases within 12 months prior to enrollment;
* Subjects who have impaired heart functions or clinically serious heart disease；
* Have severe systemic active infection;
* Have a history of tuberculosis within 1 year before enrollment, or had an active TB infection more than 1 year before but not received adequate anti-TB treatment;
* Subjects known to be allergic to the study drug or its active ingredients or excipients;
* Subjects taking known moderate or strong inducers and inhibitors of CYP3A within 14 days before the first administration;
* Active autoimmune and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic therapy, rheumatoid arthritis, inflammatory bowel disease, and Hashimoto's thyroiditis, etc., except type I diabetes, Hypothyroidism that can be controlled by replacement therapy alone, hyperthyroidism that is stable under drug control, skin diseases that do not require systemic therapy (eg, vitiligo, psoriasis);
* Past medical history of interstitial lung disease (ILD), history of drug-induced ILD, history of radiation pneumonitis requiring steroid therapy, or evidence of any clinically active ILD;
* Known impaired gastrointestinal (GI) function or GI diseases that may significantly affect the absorption or metabolism of oral drugs; abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the first administration;
* Human immunodeficiency virus (HIV) positive, syphilis (Anti-TB) positive;
* Known acute or chronic active hepatitis B (HBsAg positive or HBcAb positive, and HBV DNA ≥ 200 IU/mL or ≥ 103 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and positive for HCV RNA test);
* Subjects who experienced toxicity events during previous anti-tumor treatment and the toxicity has not resolved (the toxicity events has not been graded as ≤ level 1 according to NCI-CTCAE 5.0). Other toxicities that the investigator does not think it will affect the safety assessment of the subject (such as hair loss, etc.) will be allowed;
* Subjects who have clinically symptomatic and uncontrollable pleural or pericardial effusions after multiple times of treatments;
* Subjects who have an allogeneic tissue/ solid organ transplantation;
* Subjects who underwent major surgery within 4 weeks prior to the start of the study treatment, or who are scheduled to undergo a major surgery during the study period (procedures such as puncture or lymph node biopsy is allowed);
* Subjects who have received live vaccines (including attenuated live vaccines) within 28 days prior to the administration of study drug. Inactivated vaccines are permitted.
* A superscan as seen in the baseline bone scan；
* Subjects who are considered unsuitable for the study judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Ph Ib/IIa: Overall safety profile including adverse events | Baseline up to approximately 2 years
  Adverse Events will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version [5.0])
Ph Ib/IIa: Recommended phase 2 doses (RP2D) of XNW5004 in combination with enzalutamide | Approximately 6 months
  RP2D of XNW5004 as administered orally twice daily (BID), continuously in 28-day cycles, in combination with enzalutamide in subjects with mCRPC by safety data, pharmacokinetic data, pharmacodynamic data and efficacy data
Preliminary efficacy determination as evaluated by disease specific response criteria | Baseline until disease progression or death or through study completion (approximately 2 years)
  Radiographic Progression-free survival（rPFS）was defined as the time from the date of first administration of the study drug to the date of radiographic progression base on the investigator assessment per PCWG3 criteria or death due to any cause (whichever comes first) in Phase IIa/IIb.

SECONDARY OUTCOMES:
Ph Ib/IIa: Pharmacokinetic Parameters | The first 28-day cycle of therapy
  The area under the plasma concentration-time curve (AUC)
Ph Ib/IIa: Pharmacokinetic Parameters | The first 28-day cycle of therapy
  Maximum plasma concentration (Cmax)
Ph Ib/IIa: Pharmacokinetic Parameters | The first 28-day cycle of therapy
  Elimination half-life (t1/2)
Ph Ib/IIa: Pharmacokinetic Parameters | The first 28-day cycle of therapy
  Time to maximum plasma concentration (Tmax)
Ph Ib: Pharmacodynamic Parameters | The first 28-day cycle of therapy
  The relative change from baseline in H3K27me3 (trimethylation at lysine 27 of histone H3)/ total histone H3.
Overall Response Rate (ORR) | Baseline up to approximately 2 years
  ORR was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline reviewed by the investigator.
Disease Control Rate (DCR) | Baseline up to approximately 2 years
  DCR was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1 reviewed by the investigator.
Evaluate overall survival | Baseline up to approximately 2 years
  Overall Survival (OS) was defined as the time from the date of first administration to the date of death due to any cause.
Proportion of patients with a PSA response at week 12 | Baseline up to approximately 2 years
  Proportion of patients with a PSA response (a decrease of PSA ≥ 50% compared to baseline) after 12 weeks of treatment, which need to be confirmed more than one time consecutively by PSA test with a minimum of 3 weeks time interval.
Prostate-specific Antigen 50 (PSA50) Response | Baseline up to approximately 2 years
  Proportion of patients with a PSA response greater than or equal to 50% throughout the entire treatment course.
Time to first symptomatic skeletal event (SSE) | Baseline up to approximately 2 years
  The time from the date of the first dose of study drug to the first occurrence of a SSE, including the use of external radiation therapy (EBRT) to prevent or alleviate bone symptoms, the occurrence of new symptomatic pathological fractures (vertebrae or non vertebrae), the occurrence of spinal cord compression, and tumor related orthopaedic surgical intervention, whichever comes first.
Ph IIb：Overall safety profile including adverse events | Baseline up to approximately 2 years
  Adverse Events will be graded by National Cancer Institute Common Terminology ACriteria for Adverse Events (NCI CTCAE version [5.0])

CONTACTS AND LOCATIONS:
Overall Officials: D Ye, M.D., Principal Investigator — Dingwei Ye
Locations (2):
- China (2):
  - Cancer Hosipital of Shandong First Medical University,440 Jiyan Road, Jinan City, Shandong Province, Jinan, Shandong
  - 270 Dongan Road, Shanghai, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No